CLINICAL TRIAL: NCT00632736
Title: An Open-Label Extension Study With REQUIP (Ropinirole) CR for Subjects From Studies 101468/165, 101468/168 and 101468/169
Brief Title: An Open-label Continuation Study Evaluating the Long-term Safety of Extended Release Ropinirole XL (Formerly CR) in Parkinson''s Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101468/248
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Results first posted 2010-12-24 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease; Parkinson's Disease
Keywords: ropinirole XL; REQUIP; Parkinson's disease; long term safety; efficacy; safety; ropinirole CR; ropinirole IR; open-label
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ropinirole XL (formerly CR) (Active Comparator): Ropinirole XL (formerly CR)
  Interventions: Drug: Ropinirole XL (formerly CR)

INTERVENTIONS:
Drug: Ropinirole XL (formerly CR)

SUMMARY:
To evaluate the safety profile of ropinirole XL during long-term treatment in subjects with early and advanced Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Subjects must have completed REQUIP studies 165 or 168, or must have completed at least 12 weeks of randomised treatment in study 169 (and must have completed the one-week down titration at the end of treatment/early withdrawal).
* Subjects must not have a break in medication between completing the feeder study (including the down titration phase for studies 168 and 169) and beginning treatment in study 248.
* Women of child-bearing potential must be practicing a clinically accepted method of contraception during the study and for one month following completion of the study. Acceptable contraceptive methods include oral contraception, surgical sterilization, intrauterine device (IUD), or diaphragm IN ADDITION to spermicidal foam and condom on male partner, or systemic contraception (e.g. Norplant System).
* Provide written informed consent for this study.
* Be willing and able to comply with study procedures.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Patients with any ongoing clinically significant adverse events at the end of the "feeder" studies.
* Subjects with severe, clinically significant condition(s) other than Parkinson's disease which, in the opinion of the investigator, would render the subject unsuitable for the study (e.g., psychiatric, hematological, renal, hepatic, endocrinology, neurological (other than Parkinson's disease), cardiovascular, or active malignancy (other than basal cell carcinoma).
* Subjects with clinically significant abnormalities in Laboratory or ECG tests at the end of the feeder study (REQUIP study 165, 168 or 169).
* Subjects with severe dizziness or fainting due to postural hypotension on standing.
* Withdrawal, introduction, or change in dose of hormone replacement therapy and/or any drug known to substantially inhibit cytochrome P 450 1A2 (CYP1A2 [e.g. ciprofloxacin, fluvoxamine, cimetidine, ethinyloestradiol]) or induce CYP1A2 (e.g. tobacco, omeprazole) within 7 days prior to enrolment. Subjects already on chronic therapy with any of these agents may be enrolled but doses must have remained stable from 7 days prior to enrolment through the end of the treatment period.
* Women who are pregnant or breast-feeding.
* Use of an investigational drug throughout the treatment period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2004-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (65):
- United States (25):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Wichita Falls, Texas
  - GSK Investigational Site, Milwaukee, Wisconsin
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Hoboken
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Czechia (6):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Plzen - Lochotin
  - GSK Investigational Site, Prague
- France (3):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Rouffach
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Vasvari Pal Street 2, H=9023 Gyor
- Italy (5):
  - GSK Investigational Site, Pescara, Abruzzo
  - GSK Investigational Site, Pozzilli (IS), Molise
  - GSK Investigational Site, Grosseto, Tuscany
  - GSK Investigational Site, Lido Di Camaiore (LU), Tuscany
  - GSK Investigational Site, Vicenza, Veneto
- Poland (10):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Cibórz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Leszno
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Barcelona, Spain
- United Kingdom (5):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Chertsey, Surrey
  - GSK Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Makumi CW, Asgharian A, Ellis J, Shaikh S, Jimenez T, VanMeter S. Long-term, open-label, safety study of once-daily ropinirole extended/prolonged release in early and advanced Parkinson's disease. Int J Neurosci. 2016;126(1):30-8. doi: 10.3109/00207454.2014.991924. Epub 2014 Dec 27. PMID 25495896
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101468/248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study 101468/248 (this study, NCT00632736) was an open-label extension study with ropinirole extended release (XL) for subjects from studies 101468/165, 101468/168, and 101468/169 (NCT00381472).
Groups:
- Ropinirole XL: Ropinirole extended release (XL) doses of 8 milligrams (mg)/day, 12 mg/day, 16 mg/day, 20 mg/day, or 24 mg/day taken once daily. As this was an extension study, the dose was a continuation of the dose the participant would have been receiving in the parent study.
Period: Overall Study
Arm/Group | Ropinirole XL
Started | 419
Completed | 151
Not Completed | 268
Not completed — Adverse Event | 104
Not completed — Lost to Follow-up | 15
Not completed — Protocol Violation | 14
Not completed — Withdrawal by Subject | 99
Not completed — Lack of Efficacy | 5
Not completed — Sponsor terminated study | 5
Not completed — Non-compliance | 10
Not completed — Other | 16

BASELINE CHARACTERISTICS:
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 419
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 259
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 409
  American Hispanic | 5
  Black | 2
  Arabic/North African | 0
  East & South East Asian | 2
  South Asian | 0
  Unknown | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meters (kg/m^2)] — BMI is a measure of body fat based on height and weight and is calculated as weight (kilograms) divided by height (meters squared).
  kilograms per square meters (kg/m^2) | 26.5 (4.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Number of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs, defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, were collected to obtain data on the safety, tolerability, and benefit of ropinirole XL. SAEs, defined as AEs that are fatal, life threatening, disabling/incapacitating, resulting in hospitalization or prolongation of a hospital stay, a congenital abnormality/birth defect, or any important medical occurrence that the investigator regards as serious based on medical judgment, were also collected. st. med., study medication.
Time Frame: 13 February 2004 through 31 March 2010
Population: Safety Population: all participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 419
participants
  Participants (Par.) reporting at least one AE | 365
  Par. reporting at least one SAE | 109
  Par. with drug-related AEs | 213
  Par. with AEs leading to withdrawal | 106

2. Secondary Outcome: Number of Participants With the Indicated Response to the Patient Preference Question at Week 4 and Week 26
Description: The patient preference question assessed the participant's preference for either dosing regimen of study drug, once a day versus three times a day. Participants were asked to respond to the following question to assess preference: "Please indicate whether you preferred taking your Parkinson's tablets 3 times a day or once a day." Wk, Week.
Time Frame: Week 4 and Week 26
Population: All participants enrolled into this study from parent study 101468/168 who received at least one dose of study medication. Only 74 participants completed this questionnaire at Week 4, whereas 87 participants completed this questionnaire at Week 26.
Measure: Number; unit: participants
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 112
participants
  Very much preferred three times a day, Wk 4, n=74 | 2
  Much preferred three times a day, Week 4, n=74 | 0
  Preferred three times a day, Week 4, n=74 | 4
  Both regimens are about the same, Week 4, n=74 | 5
  Preferred once a day, Week 4, n=74 | 17
  Much preferred once a day, Week 4, n=74 | 18
  Very much preferred once a day, Week 4, n=74 | 28
  Very much preferred three times a day, Wk 26, n=87 | 4
  Much preferred three times a day, Week 26, n=87 | 1
  Preferred three times a day, Week 26, n=87 | 2
  Both regimens are about the same, Week 26, n=87 | 4
  Preferred once a day, Week 26, n=87 | 14
  Much preferred once a day, Week 26, n=87 | 20
  Very much preferred once a day, Week 26, n=87 | 42

ADVERSE EVENTS:
Arm/Group | Ropinirole XL
Serious Adverse Events (participants affected / at risk) | 109/419
Other Adverse Events (participants affected / at risk) | 261/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole XL (N=419)
Parkinson's Disease (Nervous system disorders) | 12
Dyskinesia (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 2
Akinesia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular spasm (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Hypokinesia (Nervous system disorders) | 1
Neuroleptic malignant syndrome (Nervous system disorders) | 1
Radicular syndrome (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Acute tonsillitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Post-procedural complication (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Splenic injury (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Angina pectoris (Cardiac disorders) | 5
Coronary artery disease (Cardiac disorders) | 4
Arrhythmia (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiovascular insufficiency (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Hallucination (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Hallucinations, mixed (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Death (General disorders) | 2
Chest pain (General disorders) | 1
Device breakage (General disorders) | 1
Device dislocation (General disorders) | 1
Gait disturbance (General disorders) | 1
Malaise (General disorders) | 1
Multi-organ failure (General disorders) | 1
Sudden death (General disorders) | 2
Hypertensive crisis (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary retention (Renal and urinary disorders) | 3
Bladder neck obstruction (Renal and urinary disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Ovarian cyst (Reproductive system and breast disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Blood pressure increased (Investigations) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole XL (N=419)
Somnolence (Nervous system disorders) | 47
Dyskinesia (Nervous system disorders) | 35
Headache (Nervous system disorders) | 27
Dizziness (Nervous system disorders) | 23
Parkinson's Disease (Nervous system disorders) | 23
Hallucination (Psychiatric disorders) | 54
Insomnia (Psychiatric disorders) | 31
Depression (Psychiatric disorders) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 58
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Influenza (Infections and infestations) | 23
Oedema peripheral (General disorders) | 48
Nausea (Gastrointestinal disorders) | 27
Fall (Injury, poisoning and procedural complications) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.